CLINICAL TRIAL: NCT07134491
Title: Peripheral and Intrarenal B Cell Study in Antibody Mediated Transplant Rejection : Phenotypic and Transcriptional Study, Study of Reactivity
Acronym: B-KiMi
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250908
Record Dates: First submitted 2025-07-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Antibody Mediated Rejection After Kidney Transplantation
Keywords: Kidney transplantation; Rejection; Donor-specific antibodies; Human Leukocyte Antigen; Microbiome
MeSH Terms: conditions — Rejection, Psychology | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Removal of a piece of kidney for research purposes during a biopsy or removal of the kidney as part of routine care.
  * Stool sampling
  * Additional blood sampling during care puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- kidney biopsy or graft removal for rejection: Renal transplant recipients with suspicion of rejection or undergoing kidney biopsy or graft removal
  Interventions: Biological: Piece of kidney removal; Biological: Stool collection; Biological: Blood collection
- kidney biopsy or graft removal for reasons other than rejection: Renal transplant recipients with undergoing kidney graft removal or biopsy for reansons other than rejection
  Interventions: Biological: Piece of kidney removal; Biological: Stool collection; Biological: Blood collection

INTERVENTIONS:
Biological: Piece of kidney removal — removal for a piece of kidney for research purposes during biopsy or graft removal performed as part of routine care
Biological: Stool collection — Stool collection for research purposes
Biological: Blood collection — Additional blood volume for research purposes during a routine blood collection

SUMMARY:
Humoral rejection of kidney transplants is responsible for a large number of kidney graft losses in a context of increasing shortage.

Although it has been established that it is largely mediated by the alloreactive B lymphocyte, anti-B therapies are only partially effective.

The mechanisms behind the loss of tolerance are also poorly understood, and the triggers of rejection remain to be elucidated.

During this study, patients admitted for kidney graft biopsy for suspicion of rejection will be included ; patients presenting non inflammatory biopsies will be studied as controls. B cells will be extracted and cultured. Their antibodies will be studied along with reactivity towards HLA, non HLA targets and the gut microbiome. The same study will be led for late rejections needing graft removal : B cells extraction, culture, antibodies reactivity testing. Controls will be graft removal for non inflammatory causes. In both cases hight throughput sequencing the immunoglobulin genes will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant recipients admitted for biopsy or graft removal in the participating nephrology departments.
* Patient participation agreement and signed consent form
* Affiliation to a health insurance system

Exclusion Criteria:

* Confounding factor of renal inflammation: acute or recurrent pyelonephritis, BK virus nephropathy
* Pregnant or breast-feeding women
* Persons under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study covers a population of adult kidney transplant patients admitted for biopsy or graft removal in the participating nephrology departments.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of lymphocytes in humoral rejection | Day 1
  Using Flow cytometry analysis

SECONDARY OUTCOMES:
Analyze of gut microbiota of kidney transplant patients | Day 1
  Using Flow cytometry analysis

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nephrology department, Hôpital Pitié Salpêtière, Paris
  - Nephrology department, Tenon hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.